CLINICAL TRIAL: NCT02257307
Title: Telemedicine Approaches to Evaluating Acute-Phase ROP eROP Ancillary Study - Implementation Project
Brief Title: Telemedicine Approaches to Evaluating Acute-Phase ROP eROP Implementation Project
Status: Terminated | Type: Observational
Why Stopped: expired study
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 14-010824; U10EY017014 (NIH)
Record Dates: First submitted 2014-10-02; First posted 2014-10-06 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Retinopathy of Prematurity
Keywords: ROP; retinopathy; Referral warranted retinopathy
MeSH Terms: conditions — Retinopathy of Prematurity; Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: RetCam retinal imaging used for routine care — De-identified digital images of both eyes, obtained by a non-physician Certified ROP Imager (CRI) using the RetCam Shuttle, will be uploaded to the secure server for remote evaluation by a Trained Reader. The results of the Reader's evaluation will be reported to the Clinical Center.

SUMMARY:
Evaluating retinopathy of prematurity (eROP) ancillary study Implementation Project is a multi-center observational study will focus on feasibility, and relative cost-effectiveness of an retinopathy of prematurity (ROP) telemedicine evaluation system to detect eyes of at-risk babies and provide timely feedback to the examining ophthalmologist at the Clinical Center.

DETAILED DESCRIPTION:
Study Design: Observational Cohort Study Setting/Participants: Premature babies who are at high risk for ROP during their stay in the neonatal intensive care unit (NICU).

* The number of sites - 5 centers in the US
* The number and description of participants: 500 babies with birth weights of <1251g

Study Interventions and Measures:

Data from RetCam digital images obtained as part of clinical care during the routine diagnostic eye exam for ROP will be uploaded and transmitted via secure server to a central reading center. These de-identified images will be graded by Certified Image Readers. Results of image gradings will be sent back via secure web-based platform to the Clinical Center. The primary outcome measure is the turnaround time from uploading the images to feedback to the Clinical Center. The secondary outcome measure is the time required to obtain retinal images for babies scheduled for ROP examination in the NICU (relative cost-effectiveness).

ELIGIBILITY:
Inclusion Criteria:

1. Babies with birth weights of <1251g
2. Babies having clinical examinations to screen for ROP

Exclusion Criteria:

* Referral from an outside hospital for treatment of serious ROP that is performed before imaging can be obtained.
* Congenital Non-ocular Anomalies: Babies will be excluded from this study if they have a severe congenital non-ocular anomaly. Such exclusions include anencephaly, trisomy 13, trisomy 18, or severe cardiac or pulmonary abnormalities. The neonatologist caring for the baby will determine whether a particular congenital abnormality would exclude the baby from participation in this study.
* Ocular Abnormalities: Babies will be excluded from this study if they have major congenital abnormalities in one or both eyes including microphthalmos, anophthalmos, anterior segment dysgenesis, dense corneal opacity, cataract, glaucoma, chorioretinitis, optic nerve hypoplasia, and chorioretinal coloboma. Eyelid abnormalities, such as severe blepharoptosis or severe hemangioma, that would likely affect vision, would also exclude a baby from participation. Minor abnormalities that would not be expected to affect vision may not be exclusion criteria including Mittendorf dot, mild blepharoptosis, limbal dermoid, and iris coloboma.

Ages: 32 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature babies (N=500) with birth weights of <1251g who meet current ROP screening guidelines in 5 NICUs in US.
Sampling Method: Non-Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04 (Actual); Study Completion 2016-03-16 (Actual)

PRIMARY OUTCOMES:
Determine whether imaging evaluation can be achieved for each baby within 24 hours following uploading of images in order to provide timely feedback to the examining ophthalmologist. | 6 months
  Interval from uploading the images to the secure server to the time a grading report is submitted to the Clinical Center

CONTACTS AND LOCATIONS:
Overall Officials: Graham E Quinn, MD, MSCE, Study Chair — Children's Hospital of Philadelphia
Locations (5):
- United States (5):
  - Johns Hopkins University, Baltimore, Maryland
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah